CLINICAL TRIAL: NCT03938194
Title: Image-guided Robot-assisted Waterjet Ablation of the Prostate for Patients With Retention of Urine Due to Benign Prostatic Obstruction
Brief Title: Waterjet Prostate Ablation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Equipment is not available
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Hang Yee, Honorary Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE 2019.043
Record Dates: First submitted 2019-04-23; First posted 2019-05-06 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Aquablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aquablation (Experimental): Surgery of benign prostatic hyperplasia by waterjet ablation
  Interventions: Procedure: Aquablation

INTERVENTIONS:
Procedure: Aquablation — a novel minimally invasive water ablation therapy combining image guidance and robotics for the targeted and heat-free removal of prostate tissue

SUMMARY:
Introduction Men with enlarged prostates commonly experience lower urinary tract symptoms and may go on to develop complications such as acute urinary retention (AUR). Surgery is the standard treatment option required to remove the enlarged prostates and to rectify such complications.

Transurethral resection of prostate (TURP) was first performed over 80 years ago and is still regarded as the "gold standard" for the treatment of benign prostatic enlargement (BPE) in prostates between 30 and 80ml. While TURP results in an improvement in symptoms, perioperative morbidity and long-term complications can include postoperative bleeding, urinary retention, incontinence, urethral strictures, erectile dysfunction, and ejaculatory dysfunction. Aquablation, a novel minimally invasive water ablation therapy combining image guidance and robotics (AQUABEAM®, Procept BioRobotics, Redwood Shores, CA, USA) for the targeted and heatfree removal of prostate tissue is one of the efforts in the development of new technology in recent years to replicate the effectiveness of TURP and at the same time with an improved safety profile. In this study, investigators plan to evaluate the feasibility and safety of Aquablation in the management of AUR secondary to BPE.

Method 20 participants are expected in this study. After patients consent to participate in the study, they will go through Aquablation under general anaesthesia or spinal anaesthesia. The ablation is delivered by transurethral means. After the procedure, subject is expected to go home on the following day. Subject will be assessed 3 months and 6 months after the procedure. Follow-up assessment includes blood tests, prostate ultrasound and urodynamic study.

DETAILED DESCRIPTION:
Benign prostatic enlargement (BPE) is a non-malignant growth of the prostate gland that can lead to a range of lower urinary tract symptoms (LUTS), and in some cases eventually leading to retention of urine. In patients failing to wean off catheter after retention of urine due to BPE, surgical intervention is the standard treatment.

Surgical intervention options have evolved from electrosurgical resection to the use of lasers for enucleation and ablation. Transurethral resection of prostate (TURP) was first performed over 80 years ago and is still regarded as the "gold standard" for the treatment of BPE in prostates between 30 and 80ml. While TURP results in a statistically significant improvement in symptoms score and and maximum urinary flow rate (Qmax), perioperative morbidity and long-term complications can include postoperative bleeding, urinary retention, incontinence, urethral strictures, erectile dysfunction, and ejaculatory dysfunction. Aquablation, a novel minimally invasive water ablation therapy combining image guidance and robotics (AQUABEAM®, Procept BioRobotics, Redwood Shores, CA, USA) for the targeted and heat-free removal of prostate tissue is one of the efforts in the development of new technology in recent years to replicate the effectiveness of TURP and at the same time with an improved safety profile. Safety and feasibility of Aquablation in the management of benign prostatic hyperplasia (BPH) have been proven successful in both canine model and human. Since then, two other prospective non-randomized trials demonstrated that the surgical ablation of the prostate using Aquablation had achieved significant and immediate improvement of functional voiding parameters as well as symptomatic improvement. Two randomized controlled trials comparing Aquablation against TURP found that Aquablation had produced a similar improvement in LUTS as TURP, with a better side-effect profile. AQUABEAM® is currently a FDA approved equipment for the ablation of prostate tissue. It is being used in US as well as in Europe and New Zealand.

So far, all studies focused on the application of Aquablation in patients with LUTS only secondary to benign prostatic obstruction (BPO). In this study, investigators plan to evaluate the feasibility and safety of Aquablation in the management of another facet of BPH, which is retention of urine.

ELIGIBILITY:
Inclusion Criteria:

* Retention of urine refractory to medical treatment

Exclusion Criteria:

* Patients with active urinary tract infection
* Patients with bleeding disorder or on anti-coagulation
* Patients with bladder pathology including bladder stone and bladder cancer
* Patients with urethral stricture
* Patients with neurogenic bladder and/or sphincter abnormalities
* Patients with previous nonpharmacological prostate treatment,
* Prostate cancer
* Fail to give informed consent

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only men have prostate
Enrollment: 20 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Wean off Catheter | Post operation 3 days
  % success in weaning off catheter

SECONDARY OUTCOMES:
Complication rate | Post operation 30 days
  Complications rate after study intervention
International Prostate Symptom Score (IPSS) questionnaire total Score | Post operation 3 months & 6 months
  Change in total scores in International Prostate Symptom Score (ranges from 0 to 35) questionnaires
International Prostate Symptom Score (IPSS) questionnaire QoL Score | Post operation 3 months & 6 months
  Change in quality of life assessed by International Prostate Symptom Score questionnaire (ranges from 0 to 6)
International Index of Erectile Function 5 (IIEF-5) questionnaire score | Post operation 3 months & 6 months
  Change in International Index of Erectile Function 5 questionnaire score (ranges from 0 to 25)
Overactive bladder symptom score (OABSS) questionnaire total score | Post operation 3 months & 6 months
  Change in total score in Overactive Bladder Symptom Score questionnaire (ranges from 0 - 15)
Pain Score | Post operation day 1 & 3 months
  Post-treatment pain score ranges from 1 to 10
Change in urodynamic in flowrate | Post operation 3 months
  Functional outcome 1: change in urodynamic function assessed by Uroflowmetry
Change in urodynamic in cystometry | Post operation 6 months
  Functional outcome 2: change in urodynamic function assessed by cystometrogram (CMG)

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No